CLINICAL TRIAL: NCT00155922
Title: The Gene Expression Patterns in the Peripheral White Blood Cells of Type 2 Diabetic Patients, Special Relevance to Atherosclerosis
Brief Title: The Gene Expression Patterns in the Peripheral White Blood Cells of Type 2 Diabetic Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9261700953
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2006-12-14 (Estimated); Status verified 2005-09

CONDITIONS: Diabetes Mellitus, Type 2; Atherosclerosis
Keywords: Diabetes mellitus; Monocyte; Gene expression; Monocyte gene expression
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Atherosclerosis; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

SUMMARY:
The investigators hypothesize that macrophages play a crucial role in the pathogenesis of atherosclerosis in patients with type 2 diabetes mellitus (T2DM).

DETAILED DESCRIPTION:
Cardiovascular events are the leading cause of death in developed countries worldwide, including Taiwan. Type 2 diabetes mellitus (T2DM), previously considered merely as one of the risk factors, has been recently unanimously accepted to be coronary artery disease-equivalent. How T2DM may lead to accelerated atherosclerosis remains obscure.

Hyperglycemia with or without hyperinsulinemia may lead to higher oxidative stress and generalized inflammation. The oxidative stress and inflammation may play a significant role in the pathogenesis in diabetic complications, including micro- and macro-vascular complications. Macrophages together with T-lymphocytes are the earliest cell-types found in fatty-streaks, the earliest atherosclerotic lesions. Macrophages are also well known cellular mediators of oxidative stress and inflammation. Therefore, it is plausible to hypothesize that macrophages play a crucial role in the pathogenesis of atherosclerosis in patients with T2DM. In addition, the other cell types of the peripheral white blood cells (WBC), such as neutrophils, have been shown to be intimately related to acute coronary syndrome. Therefore, the study on the biology of peripheral WBCs may tell us something about the pathophysiology of diabetic macro-vascular complications.

Methods:

1. Normal control: fasting plasma glucose (FPG) less than 126 mg/dl.
2. T2DM: FPG >＝126 mg/dl.

   * Group 1 (good glycemic control): hemoglobin A1c (HbA1c) <＝ 7% in the past 6 months
   * Group 2 (poor glycemic control): HbA1c >＝ 8% in the past 6 months
3. Blood sample will be collected at baseline and after aggressive control.

ELIGIBILITY:
Inclusion Criteria:

* Normal control: fasting plasma glucose (FPG) less than 126 mg/dl.
* T2DM: FPG >＝126 mg/dl.

  * Group 1 (good glycemic control): HbA1c<＝7% in the past 6 months
  * Group 2 (poor glycemic control): HbA1c>＝8% in the past 6 months

Exclusion Criteria:

* Acute systemic diseases

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2003-11

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Shiung Yang, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan